CLINICAL TRIAL: NCT02281682
Title: Topical Ingenol Mebutate Versus 5% 5-fluorouracil Versus 5% Imiquimod Versus Photodynamic Therapy in Treatment of Actinic Keratosis: a Multi-centre Randomized Efficacy and Cost-effectiveness Study
Brief Title: IM Versus 5-FU Versus IMI Versus MAL-PDT in Treatment of Actinic Keratosis
Acronym: Akti
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL50621.068.14; 836031011 (Other Grant/Funding Number: ZonMw); 2014-003691-23 (EudraCT Number)
Record Dates: First submitted 2014-10-28; First posted 2014-11-03 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Keratosis, Actinic
Keywords: Keratosis, Actinic; Treatment Outcome; cost-effectiveness; economic evaluation; imiquimod; photodynamic therapy; topical fluorouracil; ingenol mebutate
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod; Fluorouracil; 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Imiquimod (Active Comparator): three times a week once daily during 4 consecutive weeks. Prior to treatment: curettage
  Interventions: Drug: 5-fluorouracil; Drug: Ingenol mebutate; Procedure: methylaminolevulinate photodynamic therapy
- 5-Fluorouracil (Active Comparator): during 4 (consecutive) weeks twice daily. Prior to treatment: curettage
  Interventions: Drug: Imiquimod; Drug: Ingenol mebutate; Procedure: methylaminolevulinate photodynamic therapy
- Ingenol mebutate 0.015% (Active Comparator): during 3 (consecutive) days once daily. Prior to treatment: curettage
  Interventions: Drug: Imiquimod; Drug: 5-fluorouracil; Procedure: methylaminolevulinate photodynamic therapy
- MAL-PDT (Active Comparator): methylaminolevulinate photodynamic therapy; one session. Prior to treatment: curettage
  Interventions: Drug: Imiquimod; Drug: 5-fluorouracil; Drug: Ingenol mebutate

INTERVENTIONS:
Drug: Imiquimod — three times a week once daily during 4 consecutive weeks. Prior to treatment: curettage
  Other Names: Aldara
  Arms: 5-Fluorouracil; Ingenol mebutate 0.015%; MAL-PDT
Drug: 5-fluorouracil — during 4 (consecutive) weeks twice daily. Prior to treatment: curettage
  Other Names: Efudix
  Arms: Imiquimod; Ingenol mebutate 0.015%; MAL-PDT
Drug: Ingenol mebutate — during 3 (consecutive) days once daily. Prior to treatment: curettage
  Other Names: Picato
  Arms: 5-Fluorouracil; Imiquimod; MAL-PDT
Procedure: methylaminolevulinate photodynamic therapy — methylaminolevulinate photodynamic therapy; one session. Prior to treatment: curettage
  Other Names: MAL-PDT
  Arms: 5-Fluorouracil; Imiquimod; Ingenol mebutate 0.015%

SUMMARY:
A multi-centre randomised controled single blind clinical phase IV trial with the aim to determine the most effective treatment in terms of lesion reduction, costs and patient satisfaction in treatment of actinic keratosis (AK), when comparing topical treatment with photodynamic therapy (PDT), 5% 5-fluorouracil (5-FU) cream, 5% Imiquimod (IMI) cream and ingenol mebutate (IM) gel.

DETAILED DESCRIPTION:
Skin cancer is the most common cancer in Caucasians and therefore a major public health issue. Its incidence is increasing rapidly. Actinic keratosis (AK) is the most prevalent precancerous chronic skin condition. It can transform into squamous cell carcinoma (SCC). AK's generally arise in a skin area that has diffuse precancerous damage, a phenomenon called field cancerization. Because of its precancerous character, it is advised to treat AK and herewith prevent development into SCC. The most frequently used field-directed treatments in the Netherlands are photodynamic therapy (PDT), topical 5% f-fluorouracil (5% 5-FU) and topical 5% Imiquimod (5% IMI). Lately another topical product is approved by Dutch healthcare insurances: Ingenol mebutate (IM). Up to date, which treatment the patient will receive, does not rely on evidence-based-medicine, but generally on the preference of the physician. Current national and international guidelines state no clear recommendations for the best choice of therapy. The aim of this study determine which treatment is the most effective treatment in terms of lesion reduction, costs and patient satisfaction when comparing topical treatment with photodynamic therapy (PDT), 5% 5-fluorouracil (5-FU) cream, 5% Imiquimod (IMI) cream and ingenol mebutate (IM) gel, in treatment of actinic keratosis (AK).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Fitzpatrick skintype I-IV
* Clinically confirmed diagnosis of AK
* One joint area of minimal 25 cm2 and maximal 100 cm2 of AK
* Minimum of 5 AK lesions
* AK Olsen grade I-III
* Location: head/neck area

Exclusion Criteria:

* Received any kind of treatment for AK in the past 3 months
* (non)melanoma skin cancer in target area
* Immuno-compromised status
* Use of systemic retinoid in the past 3 months
* Use of immunosuppressant drugs in the past 3 months and / or at time of treatment (such as oral glucocorticoids, cytostatic, antibodies, drug acting on immunophilins, interferon, opioids, Tumor Necrosis Factor (TNF) binding proteins, mycofenolate mofetil (MMF), biologic agents). inhalation corticosteroids / nasal corticosteroids are permitted.
* Porphyria
* Not able to give informed consent
* Allergy to study drugs or peanut/nut/soy products
* Pregnant and breastfeeding women
* Female in child bearing potential not using contraceptive measures, during and till 3 months post-treatment
* Genetic skin cancer disorders
* Not understanding Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2014-11; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
treatment succes | 12 months
  the proportion of patients with ≥75% lesion reduction in the number of AK lesions counted at baseline in the treatment area 12 months post final treatment (≥ 75% patient clearance at 12 months).

SECONDARY OUTCOMES:
treatment failure | 12 months
  proportion of participants with <75% reduction in number of AK lesions after 3 and 12 months post final treatment compared to baseline (<75% patient clearance at 3 and 12 months).
Treatment succes at 3 months post treatment | 3 months
  proportion of participants with ≥75% reduction in number of AK lesions at 3 months post final treatment (≥ 75% patient clearance at 3 months).
complete lesion clearance | 12 months
  proportion of lesions with 100% clearance in all treated patients at 3 and 12 months post final treatment.
SCC | 12 months
  Proportion of patients who develop a SCC in the treatment area during study follow-up.
side effects | 12 months
  local skin reactions reported in patient diary, visual analogue score (VAS), Patient-reported adverse events
Cosmetic outcome | 3 and 12 months
  based on a Cosmetic questionnaire, filled in on baseline, 3 + 12 months
patient satisfaction | 12 months
  Skindex-29 questionnaire (quality of life) , Actinic Keratosis Quality of Life (AKQoL) questionnaire; filled in on baseline, 3 + 12 months
treatment compliance | 3 months
  defined as the number of applied treatments as percentage of the number of prescribed treatments, based on patient diaries and weighing returned medication.
Overall decrease in AK | 3 and 12 months
  Decrease in number AK from baseline per patient, at 3 and 12 months post final treatment.
Cost-effectiveness | 12 months
  Healthcare/treatment costs
Investigator Global Improvement Indices | 3 and 12 months
  Investigator Global Improvement Indices (IGII) at 3 and 12 months post final treatment.
Number of new lesions | 3 and 12 months
  Number of new lesions at 3 and 12 months post final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Ahmady S, Jansen MHE, Nelemans PJ, Kessels JPHM, Arits AHMM, de Rooij MJM, Essers BAB, Quaedvlieg PJF, Kelleners-Smeets NWJ, Mosterd K. Risk of Invasive Cutaneous Squamous Cell Carcinoma After Different Treatments for Actinic Keratosis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2022 Jun 1;158(6):634-640. doi: 10.1001/jamadermatol.2022.1034. PMID 35475852
- [Derived] Ahmady S, Jansen MHE, Nelemans PJ, Essers BAB, Kessels JPHM, Kelleners-Smeets NWJ, Mosterd K. The Effect of Four Approaches to Treat Actinic Keratosis on the Health-Related QOL, as Assessed by the Skindex-29 and Actinic Keratosis QOL. J Invest Dermatol. 2021 Jul;141(7):1830-1832. doi: 10.1016/j.jid.2020.12.023. Epub 2021 Jan 18. No abstract available. PMID 33476658
- [Derived] Jansen MHE, Kessels JPHM, Merks I, Nelemans PJ, Kelleners-Smeets NWJ, Mosterd K, Essers BAB. A trial-based cost-effectiveness analysis of topical 5-fluorouracil vs. imiquimod vs. ingenol mebutate vs. methyl aminolaevulinate conventional photodynamic therapy for the treatment of actinic keratosis in the head and neck area performed in the Netherlands. Br J Dermatol. 2020 Oct;183(4):738-744. doi: 10.1111/bjd.18884. Epub 2020 Feb 19. PMID 31961446
- [Derived] Jansen MHE, Kessels JPHM, Nelemans PJ, Kouloubis N, Arits AHMM, van Pelt HPA, Quaedvlieg PJF, Essers BAB, Steijlen PM, Kelleners-Smeets NWJ, Mosterd K. Randomized Trial of Four Treatment Approaches for Actinic Keratosis. N Engl J Med. 2019 Mar 7;380(10):935-946. doi: 10.1056/NEJMoa1811850. PMID 30855743